CLINICAL TRIAL: NCT06158971
Title: Feasibility Study of the Microwave Ablation System for Lung Tissue Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: phenoMapper, LLC (Industry)
Collaborators: NIH/NCI - Grant award number: R01CA218357 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-001
Record Dates: First submitted 2023-07-05; First posted 2023-12-06 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Lung Neoplasm
Keywords: flexperc medical; microwave; ablation; phenoWave; phenoMapper
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Flexible Microwave Ablation (Experimental): Soft tissue ablation will be performed using the phenoWave flexible Microwave Ablation System and Accessories on lesions in the peripheral lung. The image-guided ablation procedure may utilize a combination of the radial EBUS and conebeam CT to confirm the lesion, position of the device relative to lesion and monitor the ablation progress.
  Interventions: Device: Flexible Bronchoscopic Microwave Ablation

INTERVENTIONS:
Device: Flexible Bronchoscopic Microwave Ablation — The phenoWave flexible microwave ablation system will be used to perform soft tissue ablation in the lungs under image guidance.

SUMMARY:
Evaluation of safety and technical feasibility of the phenoWave MW Ablation System for microwave ablation of lesions in the lung.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, single-center, study to evaluate the safety and technical feasibility of using the phenoWave MW Ablation System to deliver microwave energy for ablation of lesions in the lung.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-77 years at screening.
* Confirmed NSCLC or solitary metastatic (oligometastatic) or pulmonary metastases from an extra thoracic primary tumor lung nodule through diagnostic biopsy
* Must be eligible for curative lung resection (lobectomy).
* For primary tumor, pre-ablated parenchymal tumor/lesion size ≥ 20 mm if NSCLC, or ≥ 10 mm for metastatic disease in diameter as measured from pre-operative CT image.
* Willing to participate in all aspects of study protocol for duration of study.
* Able to understand study requirements.
* Signs informed consent form.
* Boundary of tumor is at least 15 mm away from the pleura wall and/or fissure.

Exclusion Criteria:

* Any contraindication to bronchoscopy, for example:

  * Untreatable life-threatening arrhythmias.
  * Inability to adequately oxygenate the patient during the procedure.
  * Acute respiratory failure with hypercapnia (unless the patient is intubated and ventilated).
  * Recent myocardial infarction.
  * Uncorrectable coagulopathy.
* Known coagulopathy.
* Platelet dysfunction or platelet count < 100 x 109 cells/L OR taking anticoagulant or antiplatelet agents that cannot be safely ceased in the opinion of the pulmonologist or surgeon.
* History of major bleeding with bronchoscopy.
* Suspected pulmonary hypertension.
* Moderate-to-severe pulmonary fibrosis.
* Severe emphysema (GOLD III/IV) or chronic obstructive pulmonary disease (COPD) within 3cm of tumor/lesion boundary: prior COPD assessment data is evaluated and PI consent is required.
* Bullae >5 centimeter (cm) located in vicinity of target tumor/lesion.
* Any other severe or life-threatening comorbidity that could increase the risk of bronchoscopic MWA, for example:

  * American Society of Anesthesiologists (ASA) physical status classification >P3
  * Stage 3 heart failure
  * Severe cachexia
  * Severe respiratory insufficiency or hypoxia
* Ongoing systemic infection.
* Contraindication to general anesthesia.
* Inability to stop anticoagulants (e.g., heparin, Warfarin) or antiplatelet agents (e.g. aspirin, clopidogrel) prior to procedure.
* Participation in any other study in last 30 days.
* Breastfeeding women or females of childbearing potential with a positive pregnancy test prior to the procedure or the intent to become pregnant during the study.
* Life expectancy of less than 6 months.
* Prior radiation therapy treatment in the target lobe.
* Implantable pacemaker or defibrillator.

Ages: 45 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety - AE occurrence | up to 7 days post ablation
  Incidence of complications and occurrence of Adverse Events (AEs)
Safety - AE frequency | up to 7 days post ablation
  Frequency of AEs
Safety - ablated tissue assessment | up to 7 days post ablation
  Percentage of ablated tissue within tumor boundary as assessed on gross and/or histologic evaluation
Technical Feasibility | up to 7 days post ablation
  Evidence of thermal ablation in portion of the tumor as assessed on histopathology

SECONDARY OUTCOMES:
Navigational Success | Immediately after completion of procedure (day 0)
  Measured distance of phenoWave device tip relative to the planned position from CT data
Procedural Measures | Immediately after completion of procedure and navigation to the target (day 0)
  Total procedure time and navigation time to position the device

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinfort, MBBS, BMedSci, FRACP, PhD, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No